CLINICAL TRIAL: NCT02451111
Title: Rituximab With or Without Ibrutinib for Untreated Patients With Advanced Follicular Lymphoma in Need of Therapy. A Randomized, Double-blinded, SAKK and NLG Collaborative Phase II Trial.
Brief Title: Rituximab With or Without Ibrutinib for Patients With Advanced Follicular Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The premature termination is based on the decision by the SAKK board on November 14, 2020 due to the lack of further financial support for the follow up period.
Sponsor: Swiss Cancer Institute (Other)
Collaborators: Nordic Lymphoma Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAKK 35/14; 2015-001487-19 (EudraCT Number); SNCTP000001327 (Other: SNCTP)
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Follicular Lymphoma
Keywords: Rituximab; Ibrutinib; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — ibrutinib; Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab/Ibrutinib (Active Comparator): Ibrutinib capsules for 24 months (104 weeks) daily (always at the same time) in a dose of 560 mg (4 x 140 mg capsules)
  Interventions: Drug: Ibrutinib; Drug: Rituximab
- Rituximab/Placebo (Placebo Comparator): Placebo as comparator for 24 months (4 capsules daily always at the same time)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Ibrutinib — Patients will be instructed by the Investigator to take the amount of 560 mg Ibrutinib/Placebo (4 x 140 mg capsules) orally once daily with a glass of water at approximately the same time every day.
  Other Names: Imbruvica®
  Arms: Rituximab/Ibrutinib
Drug: Rituximab — Rituximab 375 mg/m2 has to be administered i.v. for the first four (4) infusions in all patients. After i.v. administration of Rituximab for the induction therapy, the administration mode can be changed to s.c. (1400 mg) in the maintenance phase dependent on the local standard of care.
  Other Names: MabThera®

SUMMARY:
Follicular lymphomas FL has been traditionally approached either by an initial watch and wait policy in the asymptomatic patient, or with single agent treatments with the purpose of maintaining a good quality of life for a prolonged time.The combination of rituximab and ibrutinib has been tested in clinical trials and appeared to be well tolerated and active. Since ibrutinib seems to achieve better results when administered for prolonged time as shown in CLL, the investigators have chosen to compare its combination with rituximab to the prolonged rituximab-only schedule that was already shown to be very active in the SAKK 35/03 trial.

The aim of the study is to investigate the efficacy, safety and tolerability of the treatment combination of Ibrutinib and Rituximab for patients with advanced follicular lymphoma in need of therapy.

DETAILED DESCRIPTION:
Follicular lymphomas FL has been traditionally approached either by an initial watch and wait policy in the asymptomatic patient, or with single agent treatments with the purpose of maintaining a good quality of life for a prolonged time.

During the last decades, treatment strategies have changed due to the continuous development and introduction of novel therapeutic approaches (including immunotherapy with interferon-alpha or monoclonal antibodies, the combination of immunotherapy with chemotherapy, and radioimmunotherapy with radiolabeled monoclonal antibodies).

For the asymptomatic patients with advanced-stage, but low tumor burden, randomized studies have confirmed that systemic treatment can be deferred until development of symptoms or organ failure (which generally occurred within 2-3 years from diagnosis) without any overall survival impairment and a watchful waiting policy has long remained a widely accepted approach.

For the symptomatic patients with more advanced tumor burden, in need of initial treatment, the combination of rituximab and chemotherapy, possibly followed by rituximab maintenance became a new standard in many countries.

In this setting of a chemotherapy-free strategy, the clinical study of rituximab combinations with other immunotherapies or with novel targeted agents is obvious relevant. Promising results have also been reported with the combination of rituximab and lenalidomide.

The combination of rituximab and ibrutinib has been tested in clinical trials and appeared to be well tolerated and active. Since ibrutinib seems to achieve better results when administered for prolonged time as shown in CLL, the investigators have chosen to compare its combination with rituximab to the prolonged rituximab-only schedule that was already shown to be very active in the SAKK 35/03 trial.

SAKK has a long tradition in treatment of FL patients with chemotherapy-free treatment based on rituximab. This is a worldwide special situation, which creates cooperation between important partners for clinical trials in this area.

The aim of the study is to investigate the efficacy, safety and tolerability of the treatment combination of Ibrutinib and Rituximab for patients with advanced follicular lymphoma in need of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP guidelines
* Histologically confirmed FL CD20+; grade 1, 2, 3a; stage III+IV; stage II not suitable for radiotherapy; all FLIPI
* Tumor specimens (slides or block) available for pathological review
* In need of systemic therapy (at least one of the following indications must be fulfilled):

  * Symptomatic disease
  * Bulky disease (≥ 6 cm)
  * Steady, clinically significant progression over at least 3 months of any tumor lesion
  * B-symptoms (weight loss > 10% in 6 months, drenching night sweats, fever > 38°C not due to infection)
  * Anemia (hemoglobin < 100 g/L) or thrombocytopenia (platelets 50-100 x 109/L) due to lymphoma
* At least one two-dimensionally measurable lesion with a longest diameter (LDi) ≥ 15 mm in contrast-enhanced 18F-FDG PET/CT* scan
* FDG-avid tumor lesion in contrast-enhanced 18F-FDG PET/CT* scan
* Age 18-85 years
* WHO performance status 0-2
* Adequate bone marrow function:

  * Absolute neutrophil count (ANC) > 1.0 x 109/L independent of growth factor support
  * Platelets ≥ 100 x 109/L or ≥ 50 x 109/L if bone marrow involvement independent of transfusion support in either situation
* Adequate hepatic function:

  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
* Adequate renal function:

  • Serum creatinine ≤ 2 x ULN and corrected calculated creatinine clearance ≥ 40 mL/min/1.73m2.
* Women of childbearing potential have a negative serum (beta-human chorionic gonadotropin) or urine pregnancy test at Screening.
* Patient compliance and geographic proximity allow proper staging and follow-up.

Exclusion Criteria:

* Tumor bulk requiring fast response
* Known central nervous system lymphoma
* Previous systemic FL therapies
* Major surgery 4 weeks prior to randomization
* Previous or concomitant malignancy diagnosed within 3 years with the exception of adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer
* History of stroke or intracranial hemorrhage within 6 months prior to randomization
* Clinically significant cardiovascular diseases such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* Known history of human immunodeficiency virus (HIV) or active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (i.v.) antibiotics
* Concomitant diseases that require anticoagulation with warfarin or equivalent vitamin K antagonists (eg. phenprocoumon), factor Xa inhibitors (e.g. rivaroxaban, apixaban), direct thrombin inhibitors (e.g. dabigatran) or platelet inhibitors/antiplatelet agents. Aspirin is allowed (up to 300 mg/d).
* Concomitant diseases that require treatment with strong or moderate CYP3A inhibitors (see http://medicine.iupui.edu/clinpharm/ddis/clinical-table/)
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved product information or known hypersensitivity to trial drugs
* Concurrent treatment with other experimental drugs or other anticancer therapy, treatment in a clinical trial within 30 days prior to trial entry
* Vaccinated with live, attenuated vaccines 4 weeks prior to randomization
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of Ibrutinib capsules, or put the study outcomes at undue risk
* Psychiatric disorder precluding understanding information of trial related topics, giving informed consent or interfering with compliance for oral drug intake
* Women who are pregnant or breastfeeding
* Patients regularly taking corticosteroids during the last 4 weeks, unless administered at a dose equivalent to Prednisone ≤ 15 mg/day for indications other than lymphoma or lymphoma-related symptoms

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
CR at 24 months determined by PET/CT scan by the IRR panel | at 24 months
  The evaluation of CR is outlined according to Cheson Criteria.. Any assessment within a window of week 102 to week 118 (inclusive) will be considered as the 24 months response assessment for determining the CR status. In addition, the CR status will be determined as follows for these specific cases:

SECONDARY OUTCOMES:
CR at 30 months determined by PET/CT scan by the IRR panel | at 30 months
MRD evaluation | baseline and week 106
  MRD evaluation will be performed using real-time PCR (polymerase chain reaction) based methods in peripheral blood and bone marrow at baseline and week 106. The proportion of patients achieving MRD negativity will be calculated for each time point of interest.
Overall response (OR) | at 24 weeks
  OR is defined as either:
  * the disappearance of all evidence of disease (CR)
  * the regression of measurable disease with no new sites (PR)
Duration of complete response (DUR) | at 12 or 24 weeks or thereafter
  The duration of CR will be calculated from when the criteria for CR are met, until documentation of relapse thereafter. Only patients with a CR will be included in this analysis.
Progression-free survival (PFS) (PFS) | at 12 or 24 weeks or thereafter
  PFS will be calculated from randomization until the first event of interest:
  * disease progression or relapse according to criteria of Cheson et al. 2014
  * death from any cause
Event-free survival (EFS) | 12, 24 or 52 weeks
  Event-free survival (time to treatment failure) will be calculated from randomization to premature discontinuation of trial treatment for any reason (e.g., insufficient response at first or second restaging at 12 or 24 weeks or at the third assessment at 52 weeks, disease progression, toxicity, patient preference, initiation of new treatment without documented progression, secondary malignancy or death).
Time to next anti-lymphoma therapy (TTNT) | at 12 or 24 weeks or thereafter
  This will be calculated from randomization until the start of the first off-trial anti-lymphoma treatment. Patients not receiving any off-trial anti-lymphoma treatment will be censored at the last follow-up visit.
Adverse Events (AEs) | record throughout treatment phase (until 30 days after last drug administration)
  AEs will be evaluated using the NCI CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Zucca, Prof, Study Chair — Oncology Institute of Southern Switzerland IOSI, Bellinzona; Bjørn Østenstad, MD, Study Chair — Oslo University Hospital; Björn Wahlin, MD, Study Chair — Karolinska University Hospital, Stockholm
Locations (42):
- Akademisches Lehrkrankenhaus Feldkirch, Feldkirch, Austria
- Denmark (4):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense Universitetshospital, Odense C
- Finland (4):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - University Hospital Tampere Radius, Tampere
  - Turku University Hospital, Turku
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - Universitetssykehuset i Nord-Norge, Tromsø
- Sweden (6):
  - Sunderby Hospital, Luleå
  - Skanes Universitetssjukhus, Lund
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Solna
  - Karolinska University Hospital, Stockholm
  - University Hospital of Umeå, Umeå
- Switzerland (23):
  - Hirslanden Klinik Aarau, Aarau
  - Kantonspital Aarau, Aarau
  - Zuger Kantonsspital, Baar
  - Kantonsspital Baden, Baden
  - St. Claraspital AG, Basel
  - Universitaetsspital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital, Bern, Bern
  - Spitalzentrum Oberwallis - Brig, Brig
  - Kantonsspital Bruderholz, Bruderholz
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre de Chimiothérapie Anti-Cancéreuse SA (CCAC), Lausanne
  - Kantonsspital Baselland, Liestal
  - Kantonsspital Luzern, Luzerne
  - Spital Thurgau (Kantonsspital Münserlingen und Frauenfeld), Münsterlingen
  - Kantonsspital Olten, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Hôpital du Valais - CHCVR, Sion
  - Spital STS AG, Thun
  - Kantonsspital Winterthur, Winterthur
  - Stadtspital Triemli, Zurich
  - UniversitätsSpital Zürich, Zurich
  - Onkozentrum Hirslanden, Zurich

IPD SHARING:
Plan to Share IPD: No